CLINICAL TRIAL: NCT00106665
Title: Intensive Care Unit(ICU)-Acquired Paresis and the Risk for Mortality and Recurrent ICU Admission (Weakness and ICU Readmission Evaluation-WIRE)
Brief Title: New Onset Weakness in Critically Ill Patients and the Risk of Death and Recurrent ICU Admission
Status: Completed | Type: Observational
Sponsor: Naeem Ali, MD (Other)
Responsible Party: Sponsor-Investigator, Naeem Ali, MD, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2004H0255
Record Dates: First submitted 2005-03-28; First posted 2005-03-29 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Muscle Weakness; Critical Illness
Keywords: ICU acquired weakness; Critical care polyneuropathy; Critical care myopathy
MeSH Terms: conditions — Muscle Weakness; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study seeks to define the morbidity of critical care polyneuropathy and to confirm that this diagnosis is, in fact, independently associated with increased mortality. Secondary information regarding the reasons for ICU readmission in patients with weakness may help in formulating cogent discharge strategies for these patients. Measurement of weakness using handgrip strength may provide a useful surrogate marker for weakness that may be more easily and uniformly applied.

Primary hypothesis:

* The development of ICU-associated weakness is independently associated with excess attributable mortality.

Secondary hypothesis:

* The development of ICU-associated weakness is associated with an increased need for ICU readmission.
* Readmission to the ICU will be a result of the development of recurrent respiratory failure or insufficiency
* Handgrip strength testing will detect ICU-associated weakness with an equivalent sensitivity as the comprehensive bedside muscle strength exam.

DETAILED DESCRIPTION:
Study Overview: This study will enroll patients requiring prolonged mechanical ventilation to identify the presence of newly acquired weakness in the ICU. Eligible patients are those that require the use of mechanical ventilation for greater than or equal to five days, because this is a significant risk factor for weakness. These patients will be enrolled and followed to detect the true relative mortality between weak and strong patients in the ICU.

To identify patients with relevant and significant weakness, this study identifies weakness in patients who survive and return to a state of normal consciousness. As such these patients, once enrolled, need to be screened daily for awakening. Once awake an assessment of peripheral muscle strength will be performed with a standard bedside neuromuscular exam and handgrip manometry.

Initial Data Collection: After consent, demographic information and risk factors for neuromuscular disease for each patient will be recorded. Blood pressure values and other data regarding the subjects' severity of illness will be collected. Any previous use of medicines during the current hospitalization that are associated with the development of weakness will be collected as well. Also any previous history of other chronic disease known to be associated with weakness (e.g. diabetes, immune system deficiency, end-stage liver disease or kidney disease) will be noted.

Screen for awakening (SA):Once daily the patient will be assessed for awakening using a standard (RASS). When the patient awake and able to follow commands they will be assessed for muscle strength exam.

Medical Research Council Strength Exam:The examiner will perform their exam on the first day that the patient is eligible by RASS screening. This same examiner will return at least twenty hours, but no more than forty-eight hours later to perform a repeat exam. The exam will be based on the Medical Research Council standard exam. Functions assessed:Upper extremity: wrist flexion, arm flexion, shoulder abduction. Lower extremity: ankle dorsiflexion, knee extension and hip flexion. Handgrip assessment: On the same day as the MRC exam the patient will be asked to perform a handgrip maneuver using the Jamar® handgrip manometer.

Clinical outcomes:

Ventilator use, Re-intubation, Recurrent ICU admission, Tracheostomy use, ICU Length of Stay and Hospital LOS

ELIGIBILITY:
Inclusion Criteria:

* Adult (age > or = 18) patients admitted to the Medical ICU
* Respiratory failure requiring mechanical ventilation > or = 5 days
* Reasonable expectation for a subsequent return of mental status

Exclusion Criteria:

* Patient's family, physician, or both not in favor of aggressive treatment of patient or presence of an advanced directive to withhold life-sustaining treatment
* Pregnancy
* Admitted to ICU from outside hospital
* New or pre-existing diagnosis causing current neuromuscular weakness
* Profound and uncorrectable hypokalemia or hypophosphatemia [K < 2.5 or P < 1.0 throughout enrollment window]
* Inability to assess muscle strength in more than six muscle groups in at least two extremities [Bilateral amputation (BKA or AKA), severe burns, skin lesions or dressings limiting ability of examiner to access and forcibly resist movement of the patients extremities]
* Inability to communicate or follow commands of the examiner [persistent coma, severe MRDD (mental retardation and developmental disabilities) or continuing necessary medication use that impairs consciousness (i.e. narcotics), non-English speaker]
* Concurrent enrollment in another clinical trial involving steroids > 20 mg/day prednisone equivalent for > 3 days, neuromuscular blockade for > 24 hours or any aminoglycosides.
* Prisoner or other subject where legal surrogate decision maker is in question

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients requireing mechanical ventilation
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2005-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | during hospitalization

SECONDARY OUTCOMES:
recurrent respiratory failure | hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Naeem A Ali, MD, Principal Investigator — Ohio State University
Locations (5):
- United States (5):
  - Indiana University Hospitals, Indianapolis, Indiana
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio

REFERENCES:
- [Derived] Ali NA, O'Brien JM Jr, Hoffmann SP, Phillips G, Garland A, Finley JC, Almoosa K, Hejal R, Wolf KM, Lemeshow S, Connors AF Jr, Marsh CB; Midwest Critical Care Consortium. Acquired weakness, handgrip strength, and mortality in critically ill patients. Am J Respir Crit Care Med. 2008 Aug 1;178(3):261-8. doi: 10.1164/rccm.200712-1829OC. Epub 2008 May 29. PMID 18511703